CLINICAL TRIAL: NCT05380700
Title: Virtual Reality Stimulation on the Intermediate Care Unit
Brief Title: Virtual Reality on the IMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK2020-00039b
Record Dates: First submitted 2022-02-21; First posted 2022-05-19 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Feasibility of Virtual Reality Stimulation for Critically Ill Patients
Keywords: Virtual Reality; Intermediate Care Unit; Critical Care; Movement Analysis

STUDY DESIGN:
Intervention Model Description: All participants receive the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Stimulation (Experimental): All participants will be receiving the standard care and additionally the VR stimulation during their stay in the intermediate care unit.
  Interventions: Device: Virtual Reality Stimulation

INTERVENTIONS:
Device: Virtual Reality Stimulation — Participants in the intervention group will be provided with up to 30 minutes of relaxing, 360-degree virtual reality (VR) stimulation and corresponding sounds, twice in 24 hours during their stay on the intermediate care unit.
  Other Names: Visuo-acoustic stimulation

SUMMARY:
The goal of this substudy (main study NCT04498585) is to determine the feasibility of applying virtual reality stimulation to patients in the intermediate care unit. Patients on this ward are generally more awake and alert than patients in the intensive care unit, thereby they are able to provide feedback about their experience. As the intermediate care unit is not without stress, examining the physiological parameters (e.g., heart rate, respiration rate, blood pressure, etc.) could also provide telling information as to the calming effect of virtual reality. The movements of these patients are also recorded using accelerometers which will provide valuable information about the characteristics of the movements that patients make while confined to their beds. These movements can act as a reference for further investigation into movements related to delirium which is a secondary outcome measure of the main study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged ≥18 years
* No severe visual or auditory impairments (strabismus, macular degeneration, retinopathy)
* German or French speaking
* Estimated length of stay (from time of study inclusion) >24 hours

Exclusion Criteria:

* Patients without calotte, with external ventricular drainage or other Intracranial pressure probes
* Patients with epilepsy
* Patients with Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of providing virtual reality stimulation | Recorded immediately after every VR stimulation
  To determine the acceptability of providing VR stimulation to patients in the intermediate care (IMC) unit based on 1) the subjective perception of the feedback, and 2) the ability of the stimulation to be maintained for minimum 20 minutes.
Safety of providing virtual reality stimulation | Safety will be determined based on the reporting of adverse or serious adverse events in the 1-hour following the completion of the VR stimulation.
  To determine the safety based on the adverse or serious adverse events reported by the medical staff, or the subjective reporting of the participant who received the VR stimulation.

SECONDARY OUTCOMES:
Heart Rate | Recorded during entire stay in the IMC (up to 24 hours)
  Changes in heart rate (beats per minute) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
Blood Pressure | Recorded during entire stay in the IMC (up to 24 hours)
  Changes in blood pressure (mmHg) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
Respiration Rate | Recorded during entire stay in the IMC (up to 24 hours)
  Changes in respiration rate (breaths per minute) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
Oxygen Saturation | Recorded during entire stay in the IMC (up to 24 hours)
  Changes in oxygen saturation (%) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.

OTHER OUTCOMES:
Movement Patterns before and after VR stimulation | Recorded during entire stay in the IMC (up to 24 hours)
  Movement patterns, measured as acceleration and rotation, will be measured using inertial measurement units. The data will be used to determine if there is a change in pattern between periods before, during, or after stimulation.
Movement Intensity before and after VR stimulation | Recorded during entire stay in the IMC (up to 24 hours)
  Movement intensity, measured as acceleration and rotation, will be measured using inertial measurement units. The data will be used to determine if there is a change in intensity between periods before, during, or after stimulation.
Cognitive Functioning | Recorded during entire stay in the IMC (up to 24 hours)
  Cognitive abilities will be measured using the Montreal Cognitive Assessment (MoCA).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hänggi, Dr. med, Principal Investigator — Department of Intensive Care Medicine, University Hospital Bern (Inelspital)
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators will ask patients to provide informed consent for sharing their anonymized data. Once the study results are published, the investigators will make the de-identified study dataset available for secondary analyses by sharing the dataset upon reasonable request.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data will be shared once study results have been published.
Access Criteria: To be determined.